CLINICAL TRIAL: NCT07089966
Title: HIV Testing Counselor-led Care to Catalyze Integration of PrEP Delivery in Family Planning Clinics: The HIV Testing Services PrEP Integration (HTS PrEP) Project
Brief Title: HIV Testing Counselor-led Care to Catalyze Integration of PrEP Delivery in Family Planning Clinics
Acronym: HTS PrEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kenneth K Mugwanya, Associate Professor: School of Medicine, Global Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00022678; R01MH136842-01 (NIH)
Record Dates: First submitted 2025-05-05; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-03

CONDITIONS: Human Immunodeficiency Virus (HIV); HIV Pre-exposure Prophylaxis
Keywords: PrEP; HIV Prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial of 20 public health clinics implementing the intervention of HTS counselor-led PrEP care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Usual care) (No Intervention): The control period (usual care) will be when the clinics are still implementing the usual care model, prior to implementing the intervention. Prior to launching the intervention, all facilities will have a baseline phase of 3 months. That time, in conjunction with other periods when the clinics are implementing usual care will serve as the control period.
- HTS counselor-led PrEP care model (Experimental): During the intervention period, all core components of PrEP delivery - including HIV testing, eligibility assessment, dispensing, adherence counseling, and provision of refills will be conducted by existing facility HTS counselor as part of standard of care.
  Interventions: Other: HTS counselor-led PrEP care model

INTERVENTIONS:
Other: HTS counselor-led PrEP care model — PrEP delivery ,including HIV testing, eligibility assessment, dispensing, adherence counseling, and provision of refills, provided by an HTS counselor
  Other Names: HTS-led PrEP
  Arms: HTS counselor-led PrEP care model

SUMMARY:
This is a cluster randomized, stepped wedge implementation study to introduce HIV testing services (HTS) counselor-led PrEP care in public health clinics in Kenya.

ELIGIBILITY:
Inclusion Criteria:

* ≥15 years of age
* Accessing health services at participating public health facilities.
* Not known to be living with HIV prior to the visit when their clinical data is first abstracted

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30000 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
PrEP screening | Up to 42 months
  Using individual client-level data at clinics, compare proportion of clients completing PrEP eligibility screening in usual care (control) versus intervention time points
PrEP initiation | Up to 42 months
  Using individual client-level data at clinics, compare PrEP initiation in usual care (control) versus intervention time points. PrEP initiation will be measured as the proportion of eligible clients starting PrEP use documented on ministry of health (MOH) tools.
PrEP continuation | Up to 42 months
  Using individual client-level data at clinics, compare PrEP continuation in usual care (control) versus intervention time points. PrEP continuation among clients initiating PrEP will be determined by clinic visit attendance and pharmacy PrEP refill records obtained by abstraction of MOH clinic records.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Mugwanya, MBChB, MS, PhD, Principal Investigator — University of Washington
Locations (2):
- Kenya (2):
  - Kenyatta National Hospital, Kisumu
  - Kenyatta National Hospital, Siaya

IPD SHARING:
Plan to Share IPD: No